CLINICAL TRIAL: NCT02494245
Title: Increasing Physical Activity in Stroke Survivors Using STARFISH, an Interactive Mobile Phone Application: a Randomised Controlled Study
Brief Title: Increasing Physical Activity in Stroke Survivors Using STARFISH, an Interactive Mobile Phone App
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Glasgow (Other)
Collaborators: Chest, Heart and Stroke Association Scotland (Other); NHS Greater Glasgow and Clyde (Other); National Heatlh Service Ayrshire and Arran (Other Government); National Health Service Lanarkshire (Unknown)
Responsible Party: Principal Investigator, Dr Lorna Paul, Reader in Rehabilitation, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STARFISH RCT
Record Dates: First submitted 2015-07-01; First posted 2015-07-10 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Stroke
Keywords: Rehabilitation; Intervention; Walking
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Active Comparator): 128 participants will take part in the STARFISH intervention
  Interventions: Other: STARFISH
- Control (No Intervention): Participants allocated to the control group will be given a booklet with general advice on physical activity.

INTERVENTIONS:
Other: STARFISH — The intervention group will take part in a four month physical activity intervention using the STARFISH app with the aim of increasing physical activity by 3000 steps per day. Participants will be provided with a smartphone for the intervention. Participants will work in groups of four but each participant will have their own individualised step count target, based on their baseline step count. If the participant reaches their step count target on at least five days of the week, then their target will be increased by 5% for the following week, up to a maximum increase of 3000 steps above baseline. Where a participant fails to reach their step count target, it remains unchanged for the following week.
  Arms: Intervention

SUMMARY:
The aim of the study is to compare physical activity in stroke survivors who have undertaken a four month physical activity intervention using the STARFISH application with a control group receiving four months of usual care.

DETAILED DESCRIPTION:
Stroke is one of the most common disabling conditions worldwide. The various physical impairments that arise from stroke may encourage a physically inactive lifestyle (Michael et al. 2005). Ninety percent of stroke survivors have some functional disability with reduced mobility being the major impairment (Gresham et al. 1975). Stroke survivors generally spend less time physically active and more time sedentary than their age-matched healthy counterparts (Alzahrani et al. 2011; Michael and Macko 2007; Rand et al. 2010) Physical inactivity following a stroke is associated with decreased muscle strength and cardiovascular fitness, decreased ability to perform activities of daily living and a heightened risk for recurrent stroke and cardiovascular disease (Ivey et al. 2005). Cardiovascular disease is the leading cause of death in chronic stroke. Inactivity and low cardiovascular fitness are two of the modifiable risk factors associated with cardiovascular disease. Activities which promote mobility and fitness are therefore vital for the prevention of further cardiovascular events.

The previous Chest, Heart and Stroke, Scotland (CHSS) funded pilot study demonstrated that community dwelling stroke survivors are significantly less physically active and spend significantly more time sedentary compared to healthy, matched controls. (Paul et al. 2015). The investigators have also reported that using the STARFISH smartphone app (described below) for six weeks had a positive effect on physical activity These pilot results support the development of a fully powered, randomised controlled trial.

Starfish description Research team members have developed STARFISH, a smartphone app, which aims to encourage users to become more physically active. The sensors within a standard smartphone record the number of steps taken per day by the individual.

STARFISH is undertaken in groups of four to facilitate social support and each group member receives a personalised daily step count target. Each person is represented by coloured fish, and participants can see their own and other group members' fish in a fish tank on their smartphone. When the participant is walking, their fish swims and blows bubbles and, as participants progress towards their daily step count target, their fish's fins and tail grow. When all group members reach their target on five days of the week, the group is rewarded by another sea creature appearing in their fish tank (e.g. a seahorse).

Aims and Objectives

The primary objective of the study is:

To compare objectively measured physical activity in community dwelling stroke survivors who have undertaken a four month physical activity intervention using the STARFISH application with a control group receiving four months of usual care.

The secondary objectives are:

1. To compare objectively measured sedentary time, activity profiles, walking endurance, walking speed, activities of daily living (ADL), fatigue, anxiety and depression, quality of life and metabolic health-risk biomarkers in community dwelling stroke survivors who have undertaken a four month physical activity intervention using the STARFISH application with a control group receiving four months of usual care.
2. To determine if the effects of the STARFISH intervention are evident two months after completion of the intervention.

Design and Methods The design is a single blind, parallel randomised control trial (RCT). An assessor, who will be blinded to the group allocation will perform the outcome measures.

Methods Participants Using pilot study data the investigators estimated that the RCT will need 58 subjects in each group to detect, with 80% power a 30% increase in step count, between intervention and control groups, at a 5% level of significance. Therefore to allow for some drop out, 128 people who fulfil the inclusion and exclusion criteria, and who give written informed consent will be recruited to the study.

Participants will be recruited through a number of routes:

* through Chest Heart & Stroke (CHSS) affiliated groups in the West of Scotland
* in NHS Lanarkshire through the stroke liaison nurses who will identify appropriate patients from stroke audit system and through the Lifestyle Group .
* in NHS Ayrshire and Arran through the physiotherapists and stroke liaison nurses
* in NHS GG&C through the Community Stroke Team Participants identified in any one of routes described above will be given a Participant Information Sheet (PIS), from the clinician or CHSS group co-ordinator. In NHS Lanarkshire potential participants identified from the database will be sent a letter and PIS from the Lead Stroke Clinician. Those interested in taking part in the study will be asked to contact the researcher using the contact details on the PIS.

Following discussion with the researcher those willing to take part will be invited to attend Glasgow Royal Infirmary (GRI) clinical research facility, NHS Lanarkshire clinical research facility and NHS Ayrshire & Arran clinical research facility . At the initial visit the participant will meet both researcher and assessor. In order to keep assessor blind to the group allocation the researcher and the assessor will see participants separately in different rooms.

Participants will see the researcher first, where they will have the opportunity to ask further questions, if they then agree to taking part in the study they will be asked to sign a consent form. Consent will also be sought to contact participant's GPs to inform them of their participation in the research study. For participants recruited from CHSS groups their GPs agreement will be sought for their participation in this study. All participants will be informed that they are free to withdraw from the study at any time.

Those who provide their informed consent will then be directed to the assessor to undergo baseline measures. All baseline measures will be made prior to group allocation, Participants will then be directed to see the researcher who will randomise them to one of the groups. The patients will be recruited in groups of 8. For the randomisation process a list of random numbers will be generated using an Excel spreadsheet. Each number will then be printed out and placed in identical, opaque envelopes, even numbers represent the Intervention group and odd numbers the Control group. Participants will be given consecutive envelopes as they are recruited so that two groups of 4 participants will be formed with each randomisation stage.

The Intervention Group:

The intervention is a four month physical activity intervention using the STARFISH app with the aim of increasing the participant's number of steps above their baseline value. Participants allocated to the intervention group will be given a mobile phone and asked to carry the phone for seven days to establish their normal level of physical activity (PA). They will work in groups of four (as explained above) but each participant will have their own individualised step count target. The initial step count target will be created by adding 10% to the mean number of steps per day recorded on the phone. At the end of each week, step counts will be reviewed from the data on the server. If the participant reaches their step count target on at least five days of the week, then their target will be increased remotely by 5% for the following week, up to a maximum increase of 3000 steps above baseline (Fitzsimons et al. 2008). Where a participant fails to reach their step count target, it remains unchanged for the following week. Participants will be notified about their step count target change via a message displayed on their smartphone screen.

Each intervention group will meet, as a group of four participants, seven days after their baseline assessment. At this visit the researcher will explain STARFISH app and provide participants with an instruction manual to refer to if needed. Initial step count targets will be calculated (as described above), agreed with participants and set. The Intervention group will then meet with the researcher 2 months later to discuss their progress, ask any questions or raise any concerns. The researcher will meet the intervention group at the end of the programme, before their second assessment (at 4 months) to collect their smartphones. At this visit a focus group, with the STARFISH group of four participants, will be undertaken to explore participants' views of the acceptability and usability of STARFISH app.

During the intervention period participants will be given contact numbers of the researcher to call if they experience any problems.

The Control Group:

Participants allocated to the control group will be given a booklet with general advice on physical activity.

All participants will be sent a lay summary of the study at the end. Outcome measures will be taken at baseline, 4 months (end of the intervention, primary end point) and 6 months (two months after the intervention).

Descriptive statistics will be used to summarise all variables at each time point. Group differences and interaction effects for each variable will be assessed using a two-factor repeated measures ANOVA model with a Greehosue-Geisser correction factor. Model assumptions will be checked and if required appropriate transformation will be used. Where a significant Time effect is found Tukey's post hoc test will be used. Effect sizes will be reported as will estimates of observed power. All analysis will be performed on IBM SPSS v22 and the level of significance will be set at 5%.

ELIGIBILITY:
Inclusion Criteria:

* single unilateral stroke
* discharged from active rehabilitation
* the ability to walk independently, with or without using an aid or orthosis
* the ability to comprehend instruction

Exclusion Criteria:

* a history of serious cardiac disease (e.g. myocardial infarction, unstable angina) in the previous six months
* uncontrolled blood pressure
* significant neurological or musculoskeletal conditions in addition to stroke
* currently participating in another clinical trial (rehabilitation or pharmacological)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2015-10 (Actual); Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Change in the mean number of steps per day | Baseline, 4 months, 6 months
  measured with an ActivPAL activity monitor (PAL Technologies, Glasgow, Scotland)

SECONDARY OUTCOMES:
Change in sedentary time | Baseline, 4 months, 6 months
  measured with ActivPAL
Change in the Six-Minute Walk Test (6MWT) | Baseline, 4 months, 6 months
  It measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they walk back and forth along a marked walkway.
change in 10-Metre Walking Test (10MWT) | Baseline, 4 months, 6 months
  The total marked distance will be 14 meters and, to allow for acceleration and deceleration, participants will be timed over the middle 10 meters. Participants will walk the distance twice and the average of 2 trials will be measured.
Change in the Nottingham Extended Activities of Daily Living Scale (EADL) | Baseline, 4 months, 6 months
  It is an instrumental ADL scale, which is a brief, easy to understand, self-administered, questionnaire.
Change in Fatigue Severity Scale (FSS) | Baseline, 4 months, 6 months
  It is a nine item questionnaire that assesses the effect of fatigue on daily living
Change in Stroke Specific Quality of Life Scale (SS-QOL) | Baseline, 4 months, 6 months
  It is a self-report questionnaire consisting of 49 items in the 12 domains of energy, family roles, language, mobility, mood, personality, self-care, social roles, thinking, upper extremity (UE) function, vision, and work/productivity. Higher scores indicate better functioning.
change in The Hospital Anxiety and Depression Scale (HADS) | Baseline, 4 months, 6 months
  It is a 14-item self-report scale that consists of two sub scales: depression and anxiety, each with 7 items. Items are rated on a 4-point scale ranging from 0 to 3, generating a scale range of 0 to 42 points, with higher scores representing greater symptom severity. Participants, who score above 8, will be advised to contact their GP before being allowed to take part in the study.
change in blood pressure | Baseline, 4 months, 6 months
  It will be taken according to the British Hypertension Society guidelines: the patient will be in a sitting position for five minutes and three readings on the unaffected side will be taken then the mean will be calculated. At the initial assessment if the result exceeds 190/100 the person will be advised to contact their GP before being allowed to take part in the study.
Change in weight in kg | Baseline, 4 months, 6 months
  measured using calibrated scale with the subject barefoot
Change in plasma lipid profile | Baseline, 4 months, 6 months
  analysis
Change in heart rate | Baseline, 4 months, 6 months
  measured using calibrated scale with the subject barefoot
Change in walking time | Baseline, 4 months, 6 months
  measured with ActivPAL
Change in walking intensity | Baseline, 4 months, 6 months
  measured with ActivPAL
liver function (ALT, AST, GGT) | Baseline, 4 months, 6 months
  analysis
Change in C-reactive protein level (CRP, a marker of inflammation) | Baseline, 4 months, 6 months
  analysis
Change in HBA1c | Baseline, 4 months, 6 months
  analysis

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - NHS Forth Valley, Falkirk
  - NHS Greater Glasgow and Clyde, Glasgow
  - NHS Lanarkshire, Glasgow
  - NHS Ayrshire &Arran, Irvine

REFERENCES:
- [Result] Michael KM, Allen JK, Macko RF. Reduced ambulatory activity after stroke: the role of balance, gait, and cardiovascular fitness. Arch Phys Med Rehabil. 2005 Aug;86(8):1552-6. doi: 10.1016/j.apmr.2004.12.026. PMID 16084807
- [Result] Gresham GE, Fitzpatrick TE, Wolf PA, McNamara PM, Kannel WB, Dawber TR. Residual disability in survivors of stroke--the Framingham study. N Engl J Med. 1975 Nov 6;293(19):954-6. doi: 10.1056/NEJM197511062931903. PMID 1178004
- [Result] Alzahrani MA, Ada L, Dean CM. Duration of physical activity is normal but frequency is reduced after stroke: an observational study. J Physiother. 2011;57(1):47-51. doi: 10.1016/S1836-9553(11)70007-8. PMID 21402330
- [Result] Michael K, Macko RF. Ambulatory activity intensity profiles, fitness, and fatigue in chronic stroke. Top Stroke Rehabil. 2007 Mar-Apr;14(2):5-12. doi: 10.1310/tsr1402-5. PMID 17517569
- [Result] Rand D, Eng JJ, Tang PF, Hung C, Jeng JS. Daily physical activity and its contribution to the health-related quality of life of ambulatory individuals with chronic stroke. Health Qual Life Outcomes. 2010 Aug 3;8:80. doi: 10.1186/1477-7525-8-80. PMID 20682071
- [Result] Ivey FM, Macko RF, Ryan AS, Hafer-Macko CE. Cardiovascular health and fitness after stroke. Top Stroke Rehabil. 2005 Winter;12(1):1-16. doi: 10.1310/GEEU-YRUY-VJ72-LEAR. PMID 15735997
- [Result] Paul L, Brewster S, Wyke S, Gill JM, Alexander G, Dybus A, Rafferty D. Physical activity profiles and sedentary behaviour in people following stroke: a cross-sectional study. Disabil Rehabil. 2016;38(4):362-7. doi: 10.3109/09638288.2015.1041615. Epub 2015 May 4. PMID 25936730
- [Result] Fitzsimons CF, Baker G, Wright A, Nimmo MA, Ward Thompson C, Lowry R, Millington C, Shaw R, Fenwick E, Ogilvie D, Inchley J, Foster CE, Mutrie N. The 'Walking for Wellbeing in the West' randomised controlled trial of a pedometer-based walking programme in combination with physical activity consultation with 12 month follow-up: rationale and study design. BMC Public Health. 2008 Jul 26;8:259. doi: 10.1186/1471-2458-8-259. PMID 18655723
- [Derived] Saunders DH, Mead GE, Fitzsimons C, Kelly P, van Wijck F, Verschuren O, Backx K, English C. Interventions for reducing sedentary behaviour in people with stroke. Cochrane Database Syst Rev. 2021 Jun 29;6(6):CD012996. doi: 10.1002/14651858.CD012996.pub2. PMID 34184251